CLINICAL TRIAL: NCT01341418
Title: Randomized Clinical Trial of Suprapatellar Versus Infrapatellar Tibial Nailing: A Pilot Study
Brief Title: Suprapatellar Versus Infrapatellar Nailing in Tibial Fractures: A Pilot Study
Acronym: SP-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Orthopaedic Institute (Network)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-2676-3103; OTA 39 (Other Grant/Funding Number: Orthopaedic Trauma Association)
Record Dates: First submitted 2011-04-20; First posted 2011-04-25 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Tibial Fractures
Keywords: tibia; suprapatellar
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suprapatellar approach (Active Comparator): surgical approach for intramedullary nailing of the tibia
  Interventions: Procedure: Suprapatellar approach
- Infrapatellar approach (Active Comparator): surgical approach for intramedullary nailing of the tibia
  Interventions: Procedure: Infrapatellar approach

INTERVENTIONS:
Procedure: Suprapatellar approach — Suprapatellar surgical approach will be used for intramedullary nailing of tibial fractures. Arthroscopic photos will be obtained before and after nail insertion. Postoperative radiographs, outcome questionnaires and an MRI will be performed over ther course of one-year follow-up.
  Other Names: semi-extended approach
  Arms: Suprapatellar approach
Procedure: Infrapatellar approach — The Infrapatellar surgical approach will be used for intramedullary nailing of tibial fractures. No arthroscopic examination for this intervention. Postoperative radiographs, outcome questionnaires and an MRI will be performed over ther course of one-year follow-up.
  Other Names: standard tibial nailing approach
  Arms: Infrapatellar approach

SUMMARY:
This study compares two techniques for the fixation of tibial fractures. The techniques are the suprapatellar (above knee)or infrapatellar (below knee) approach to tibial intramedullary nailing. Null hypothesis: There is no difference in 1) residual post-operative pain levels, 2)knee function, 3) healing and alignment of the tibia, or 4) trochlear changes in the patello-femoral cartilage between patients who are randomized to receive tibial nail insertion through either a suprapatellar nail entry portal or a standard patellar tendon approach.

DETAILED DESCRIPTION:
Patients undergoing tibial fracture repair will be consented and randomized into one of the two techniques, with arthroscopic photos taken before and after nail insertion to study the condition of the patello-femoral cartilage. Enrolled patients will be followed for one year in clinic.

ELIGIBILITY:
Inclusion Criteria:

* Tibial shaft fractures amenable and indicated for repair with intramedullary nails, with or without the use of reaming
* Acute tibial fractures within 4 weeks of injury
* Closed or open tibial fractures after appropriate irrigation and debridement
* Fractures must be within metaphyseal/diaphyseal junctures defined as middle 3/5 of tibia
* Skeletally mature patient
* Age 18 and above.

Exclusion Criteria:

* Tibial shaft fractures that require articular reconstruction with plates
* Any tibial fracture extending > 1 cm into the proximal or distal 1/5 of tibia
* Tibial plateau fractures
* Pilon fractures
* Periprosthetic fractures
* Non-unions
* Prior knee surgery
* History of gout or rheumatoid or osteoarthritis
* Concomitant injury to same limb (including any traumatic injury to ipsilateral knee, femur or foot, and knee dislocation)
* Spinal injury
* Prisoner or high likelihood of incarceration
* Not likely to follow-up in the estimation of surgeon
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2014-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
residual postoperative knee pain | 1 year
  A Visual Analog Scale (VAS) will be used for knee pain, as well as a pain location diagram and a Lysholm knee score.

SECONDARY OUTCOMES:
union/alignment of tibia | 3 months postoperatively
  AP and lateral radiographs will be used to evaluate union/alignment of the tibia.
knee function | 6 months postoperatively
  A Lysholm knee score will be used to evaluate knee function, as well as range of motion (ROM) measurements.
trochlear changes in the patello-femoral cartilage | 1 year
  Pre- and post-nailing arthroscopic photos and an MRI at 12 months postoperative will be used to evaluate trochlear changes.

CONTACTS AND LOCATIONS:
Overall Officials: Roy W Sanders, M.D., Principal Investigator — Florida Orthopaedic Institute
Locations (2):
- United States (2):
  - Tampa General Hospital, Tampa, Florida
  - St. Josephs Hospital, Tampa, Florida

REFERENCES:
- [Background] Gelbke MK, Coombs D, Powell S, DiPasquale TG. Suprapatellar versus infra-patellar intramedullary nail insertion of the tibia: a cadaveric model for comparison of patellofemoral contact pressures and forces. J Orthop Trauma. 2010 Nov;24(11):665-71. doi: 10.1097/BOT.0b013e3181f6c001. PMID 20926959